CLINICAL TRIAL: NCT03066856
Title: Lifestyle and the Penetrance of BRCA Mutation
Brief Title: Dietary Intervention and BRCA Penetrance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Collaborators: Istituto Oncologico di Bari (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 106/13
Record Dates: First submitted 2017-02-20; First posted 2017-03-01 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Dietary Modification; BRCA1 Mutation; BRCA2 Mutation; Breast Cancer
Keywords: BRCA genes; Mutation carriers; IGF-I; Diet
MeSH Terms: conditions — Breast Neoplasms | interventions — Diet Therapy

STUDY DESIGN:
Intervention Model Description: BRCA mutation carriers, with or without breast cancer, aged 18-70 years and without metastases are eligible. After the baseline examinations, women are randomized to an active dietary intervention or to a control group. The intervention group should attend six full days of activities over the next six months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): After baseline examinations, participants are randomized to an active dietary intervention group.The intervention group is invited to attend six full days of life-style intervention activities over the next six months. These activities include six cookery courses followed by lunch, six physical activity sessions (walking for 45 minutes) and six conferences. The intervention and control groups both complete questionnaires on adherence to the Mediterranean diet (MEDAS) at baseline and at the end of the study, and are asked for at least two 24-hour recalls of the previous day's food intake, and details of their physical exercise during the six-month intervention.
  Interventions: Other: Dietary intervention
- Control (No Intervention): All participants receive general recommendations for the dietary prevention of cancer. After baseline examinations, women randomized in the control group carry on following the baseline recommendations.

INTERVENTIONS:
Other: Dietary intervention — The main aim of the trial is to reduce serum levels of IGF-I and IRm with a a low- calorie and low-protein diet. In humans, calorie restriction alone does not seem to significantly lower IGF-I; protein restriction is also required. In detail, recommendations for participants included in the intervention arm include:
  * reducing protein intake, mainly milk and animal protein (except fish), down to 10-12% of total calorie intake.
  * reducing high glycemic index food and high insulinemic foods.
  * reducing sources of saturated fat (red and processed meat, milk and dairy products).
  * eating mostly food of plant origin, with a wide variety of seasonal products.
  Arms: Intervention

SUMMARY:
Insulin-like growth factor I (IGF-I) and other markers of insulin resistance (IRm) might modulate the penetrance of BRCA genes mutation.

The investigators have designed a demonstration project with BRCA mutation carriers (with or without a previous diagnosis of breast cancer) to test:

1. whether a lifestyle intervention significantly reduceIGF-I and the other IRm (randomized trial).
2. whether mutation carriers with a previous diagnosis of breast cancer have higher IRm than carriers without breast cancer (case-controlstudy).
3. whether IRm and their change over time affect subsequent breast cancer incidence and prognosis (cohort follow-up).

The investigators expect to significantly reduce IGF-I and IRm, to find that BRCA mutation carriers with a previous breast cancer have higher IRm levels, and, in the long term, that women with persistent higher IRm levels have higher penetrance and worst prognosis.

Confirming a significant reduction of IRm and the impact of their levels on prognosis would help to develop primary prevention recommendations for high risk families.

DETAILED DESCRIPTION:
Abdominal obesity and high body weight are associated with a greater risk of breast cancer (BC) in women belonging to high risk families than in women without family history of BC. A case-control study showed that high energy intake, usually associated with higher bio-availability of growth factors, is associated with BC risk in BRCA mutation carriers. A multinational case-only study on 3000 young BC women suggested that patients with BRCA mutation had higher consumption of milk. Milk directly stimulates insulin production and release, and is associated with higher plasma levels of insulin-like growth factor I (IGF-I).

In a case-control analysis on 308 high genetic risk women, investigators showed that high serum levels of IGF-I are associated with a significantly increased penetrance.

Consistently, mechanistic studies hypothesized a functional interaction between the BRCA genes and the IGF-I system.

The lifetime cumulative risk (penetrance) of BC associated with BRCA mutations is of the order of 50%, and a sizeable proportion of mutation carriers does not develop the disease. Therefore, the penetrance of the genetic trait may be regulated trough other genetic or environmental factors, including dietary, metabolic, and growth factors. The investigators hypothesized that markers of insulin resistance (IRm), such as plasma level of glucose, insulin, IGF-I and the presence of metabolic syndrome, which affect risk and prognosis of sporadic BC, are relevant also for hereditary BC.

The investigators have designed a demonstration project with BRCA mutation carriers (with or without a previous diagnosis of BC) to test:

1. whether a lifestyle intervention significantly reduce IRm (randomized trial).
2. whether mutation carriers with a previous diagnosis of BC have higher IRm than carriers without BC (case-control study).
3. whether IRm and their change over time affect subsequent BC incidence and prognosis (cohort follow-up).

In a pilot phase the investigators have randomized 150 BRCA mutated women to a dietary intervention and a control group for a short term (6 months) trial to test the reduction of IRm levels. In the present study the investigators to recruit 600 BRCA mutation carriers to test if blood levels of IRm and their change over time influence the risk of BC and of BC relapse. All participants will receive the WCRF Decalogue for the prevention of cancer. Participants will be then randomized in an active lifestyle intervention group (6 full days of life-style intervention activities along the subsequent 6 months) and in a control group that will remain with the baseline recommendation. After 6 months also the control group will be invited to an active intervention.

The investigators expect to significantly reduce IRm, to find that BRCA mutation carriers with a previous BC have higher IRm levels, and, in the long term, that women with persistent higher IRm levels have higher penetrance and worst prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Eligible study subjects are women, aged 18-70, either unaffected or affected with BC, without metastases or previous ovarian cancer, who underwent genetic counselling and fulfilled high-risk selection criteria for genetic testing based on personal and/or family history and resulted carriers of deleterious BRCA mutations.

Exclusion Criteria:

* Unaffected BRCA mutation carriers with bilateral prophylactic mastectomy are not included in the cohort or are censored at the time of surgery.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 502 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Reduction of serum levels of IGF-I (ng/mL) (intervention trial). | 6 months of dietary intervention
  Final analyses will be performed by intention to treat. By assuming that:
  a) the planned lifestyle interventions may reduce IGF-I levels by 10%, b) alpha error = 0.05, the investigators shall have 96% power to compare 300 women included in the intervention group versus 300 in the control group.
Case-control analysis: comparison of the affected versus the unaffected BRCA mutation carriers for the baseline IRm levels baseline serum levels of IGF-I and IRm. | 3 years
  By classifying the exposure status according to the IGF-I median level and by assuming that :
  1. the probability of exposure among controls is 50 %,
  2. a case/control ratio of 2/1 (as in a pilot study): 400 women with a previous diagnosis of BC and 200 unaffected,
  3. the true odds ratio for BC in exposed versus unexposed subjects ranging between 1.5 to 2 (the lower confidence interval of a pilot study), the investigators will be able to reject the null hypothesis ( that this odds ratio equals 1) with a power ranging from 64% to 97% at the alpha level of 0.05.

SECONDARY OUTCOMES:
Survival analysis: evaluation of the association between IGF-I and IGF-I changes and subsequent BC incidence and BC prognosis (BC incidence for unaffected women and ipsilateral or contralateral BC and BC recurrences for affected women). | 3 years
  This secondary aim requires the follow-up of the BRCA mutation carriers cohort. By assuming : a) equal number of exposed (IGF-I level>median) and unexposed subjects of 300, b) 85% probability of event-free after 48 months of follow-up c) the true hazard ratio of exposed subjects relative to unexposed subjects ranging between 1.5 to 2, the investigators will be able to reject the null hypothesis that exposed and unexposed survival curves are equal with a power ranging from 41% to 78% at the alpha level of 0.05. Further follow-up will increase the power.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Italy

IPD SHARING:
Plan to Share IPD: No
Individual participant data are not available to other researchers. The data software is blinded and protected.

REFERENCES:
- [Derived] Bruno E, Oliverio A, Paradiso A, Daniele A, Tommasi S, Terribile DA, Filippone A, Digennaro M, Pilato B, Danza K, Guarino D, Rossi C, Rossi MM, Venturelli E, Giussani M, Peissel B, Pasanisi P. Lifestyle Characteristics in Women Carriers of BRCA Mutations: Results From an Italian Trial Cohort. Clin Breast Cancer. 2021 Jun;21(3):e168-e176. doi: 10.1016/j.clbc.2020.11.002. Epub 2020 Nov 10. PMID 33357965